CLINICAL TRIAL: NCT05087277
Title: Study on the Correlation of Isotype Switching, Neutralizing Antibody Titer and Cross Immunity Against COVID-19 Variants After Primary and Booster Vaccination
Brief Title: Correlation Study of Isotype Switching and Neutralizing Capacity to the COVID-19 Variants Strain
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centers for Disease Control and Prevention, China (Other Government)
Responsible Party: Principal Investigator, Wu Jiang, Director of Institute for Vaccines and Immunization, Centers for Disease Control and Prevention, China
Other Study IDs: BJCDCWJ202102
Record Dates: First submitted 2021-10-19; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: COVID-19
Keywords: cohort study; Isotype Switching; Neutralize antibodies; COVID-19 Variants Strain
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The level of neutralizing antibody was detected by using the constructed pseudovirus covid-19 variant at baseline , 1 month , 6 months and 12 months after primary vaccination, within 15 days after booster immunization at 12 months . and the ability of IgG subclasses to neutralize and cross immunization of variant strains was analyzed.

DETAILED DESCRIPTION:
In 150 individuals who received primary and booster COVID-19 inactivated vaccine, the neutralization ability of antibodies against covid-19 mutant after primary and booster immunization was evaluated by constructing pseudotyped SARS-CoV-2 variants. The contribution and influence of IgG subclasses on neutralization capacity were assessed by Elisa assay. All participants were recruited aged between 18 and 59 years old. Every participant was familiarized with the aim of the study and asked to sign an informed consent agreement and was required blood sampling at the day 0 of first dose vaccine and 1 month, 6 months after 2nd dose of primary immunization. All participants had received 1 dose of booster immunization at 12 months after fully primary vaccination. Then 150 people were divided into four groups, Blood samples were taken on days 0,3,7,10 and 14 to detect neutralizing antibodies and IgG subclasses separately. every sample was detected SARS-CoV-2 variants strain Alpha, Beta and Delta neutralizing antibody, and RBD-IgG1, IgG2, IgG3, and IgG4. every individual was conducted a detailed analysis correlation of isotype switching, neutralizing antibody titer and cross immunity against COVID-19 variants after primary and booster vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 59
* Healthy
* No vaccination with COVID-19 before become participant
* Agreed to take a blood sample

Exclusion Criteria:

* who cannot take the COVID-19 vaccine due to some personal reasons
* history of SARS-CoV, SARS-CoV-2, or Middle East respiratory syndrome infection
* high-risk epidemiology history within 14 days before enrolment (eg, travel or residence history in communities with case reports, or contact history with someone infected with SARS-CoV-2)
* axillary temperature of more than 37·0℃
* history of allergy to any vaccine component.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The healthy people aged between 18 and 59, and have not been infected with COVID-19, have not been vaccinated with COVID-19 vaccine, and agree to collect blood samples.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2021-10-10 (Actual); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
Neutralizing capabilities to variant COVID-19 after primary and booster vaccination | Baseline，After fully vaccinated 1 and 6 months，Within 15 days after booster immunization at 12 months
  The titers of neutralizing antibodies against live SARS-CoV-2 and Pseudotyped SARS-CoV-2 Variants strain Alpha, Beta and Delta at baseline, after fully vaccinated 1 and 6 months and Within 15 days after booster immunization at 12 months.
  The neutralizing antibodies was defined as a change from seronegative at baseline to seropositive or a four-fold titer increase. The positive cutoff of the titer for neutralizing antibodies was 1/30.
Titer of Subclass of IgG after primary and booster vaccination | Baseline，After fully vaccinated 1 and 6 months，Within 15 days after booster immunization at an interval of 12 months
  The titers of Subclass RBD-specific IgG1, IgG2,IgG3 and IgG4 at baseline, after fully vaccinated 1 and 6 months and Within 15 days after booster immunization at an interval of 12 months. The positive for IgG1, IgG2,IgG3 and IgG4 antibodies are defined as the sample titer value ≥1/20.

SECONDARY OUTCOMES:
Titer of subclass of IgG at different points in time after booster vaccination | 0,3,7,10,14 days
  Titer of subclass of IgG at 0,3,7,10,14 days after booster vaccination. The positive for IgG1, IgG2,IgG3 and IgG4 antibodies are defined as the sample titer value ≥1/20.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Disease Control and Prevention, Beijing, China